CLINICAL TRIAL: NCT05336097
Title: Minder Stress en Armoede, Meer Ervaren Gezondheid en Participatie
Brief Title: Pathways to Empowerment for Persons Living in Persistent Poverty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Movisie (Unknown); Municipality of Meppel, the Netherlands (Unknown); Municipality of Midden-Groningen, the Netherlands (Unknown); Municipality of Nieuwegein, the Netherlands (Unknown); Municipality of Nijmegen, the Netherlands (Unknown); Municipality of Oss, the Netherlands (Unknown); Stichting Lezen en Schrijven (Unknown); Vereniging Valente (Unknown); Voedselbanken Nederland (Unknown); Wageningen University and Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: R0005311; NWA.1239.18.003 (Other Grant/Funding Number: NWO)
Record Dates: First submitted 2022-04-05; First posted 2022-04-20 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Perceived Stress; Persistent Poverty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): Participants will receive support from participation coaches trained in Pathways to Empowerment (PTE).
  These participation coaches received a four-day training program with two weeks in between each training day, allowing them to immediately implement their acquired set of knowledge and skills. At the end of the training program, participation coaches had to successfully pass an end assignment to become PTE-certified.
  In order to ensure the implementation of PTE, the training will be supplemented with a learning cycle. This cycle consists of two workshops on poverty and stress, and of on-the-job coaching. The coaching is tailored to the wishes and needs of the team.
  Interventions: Other: Pathways to Empowerment

INTERVENTIONS:
Other: Pathways to Empowerment — Pathways to Empowerment (PTE) is a program for person-centered intervention. PTE is rooted in the Strengths Model by Rapp and Goscha (2011), and in the Social Quality Approach as described by Van der Maesen and Walker (2005). The general aim of PTE is to improve the quality of the daily lives of persons who experience loss of control in their lives by focusing on their strengths and stimulating their personal agency, participation in society, and self-direction in life. The main task of professionals is to help create the conditions in which growth and recovery are likely to occur.
  Other Names: Krachtwerk

SUMMARY:
The general purpose of this feasibility study is to evaluate the potential impact of Pathways to Empowerment (PTE) on the four constitutional conditions of social quality for persons living in persistent poverty. PTE is a strengths-based methodology developed for social care professionals to support persons in vulnerable positions with their recovery. PTE was chosen for evaluation based on in-depth interviews about appropriate support, a literature search, and participatory action research in which the wishes of each participating municipality were explored.

DETAILED DESCRIPTION:
This study is conducted with a team of participation coaches in the municipality of Nijmegen, the Netherlands. Participation coaches guide long-term recipients of social assistance benefits to a form of participation (e.g., volunteer work, sport activities, (language) courses). The team of participation coaches will be trained in PTE and will recruit participants for this study.

Participants are persons living in persistent poverty who started a support trajectory with a participation coach. Participation coaches will conduct personal conversations with potential participants, during which they will explain what this study entails, and will hand them an information letter. When potential participants express interest in participation, an interviewer will contact them by phone to provide more information about the study, to answer any questions and to schedule an interview.

Data will be collected using computer-assisted personal interviews (CAPI). These interviews will mainly be conducted by video conferencing, although participants can also be interviewed by phone or in person if they prefer. Participants are interviewed at the start of their professional support trajectory, and six months later.

At the start and at follow-up, survey data will be collected on participants' outcomes in various domains. In addition, a third semi-structured interview will be conducted with clients about their experiences with and the experienced impact of the professional support they received. This interview will be conducted around the same time as the follow-up survey, unless the provision of professional support stops before this moment. In that case, this interview is planned as soon as the participation coaches notify the research team of ending the support trajectory. Furthermore, a survey and a semi-structured interview will be conducted among participation coaches and the team manager to map their individual and job characteristics (e.g., years of working experience, caseload), and gain insight into model fidelity of PTE.

All data will be stored on secured servers of Radboudumc, for a period of 15 years. Only researchers affiliated with this project will have access to these data.

Note: Originally, two service settings participated in the study: (1) three teams of ambulatory care workers of an organization called 'Santé Partners', situated in the municipalities of Nieuwegein, Houten and IJsselstein, the Netherlands; and (2) one team of participation coaches employed at the municipality of Nijmegen, the Netherlands. The study design was altered in two crucial ways: In the first service setting, the study was terminated, and in the second service setting, the design was changed to a feasibility study and supplemented with a qualitative impact assessment.

In the first setting, ambulatory care workers in the intervention group did not take on new (eligible) clients during the recruitment period due to staff shortage. Later, the team was disbanded, as they did not receive next year's tender. Despite efforts of the researchers, it turned out to be impossible to find a substitute for this team. The study was consequently terminated in this setting.

In the second setting, the recruitment of participants by participation coaches was slower than expected. The study design was therefore changed to a feasibility study. The survey was shortened, and the quantitative data were supplemented with a qualitative evaluation of the impact of professional support based on PTE. In addition, to increase the number of participants, the recruitment period was extended. As a result, the time between baseline and follow-up was shortened from seven to six months.

ELIGIBILITY:
Inclusion Criteria:

* Participants are 18 years of age or older;
* Participants started a support trajectory at one of the participating teams during the recruitment period;
* Participants are living in persistent poverty. This means that participants have been having insufficient means for minimum living expenses and social participation for at least three years.

Exclusion Criteria:

* Being unable to provide reliable answers (e.g., having a psychotic episode);
* No informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2023-07-10 (Actual); Study Completion 2023-07-10 (Actual)

PRIMARY OUTCOMES:
Change in score on Perceived Stress Scale (PSS) | Baseline, 9 months (area of Nieuwegein) or 7 months (area of Nijmegen)
  The PSS is a 10-item instrument that measures frequency of thoughts and feelings related to perceived stress. Answers are expressed on a scale ranging from (0) "never" to (4) "very often". The PSS has been validated and widely used in the general population.

SECONDARY OUTCOMES:
Change in score on Mental Health Inventory 5 (MHI-5) | Baseline, 9 months (area of Nieuwegein) or 7 months (area of Nijmegen)
  MHI-5 is a 5-item instrument that measures mental health status. The instrument includes items on (1) anxiety, (2) general positive affect, (3) depression, and (4) behavioral/emotional control.
Change in score on Pearlin Mastery Scale (PMS) | Baseline, 9 months (area of Nieuwegein) or 7 months (area of Nijmegen)
  The PMS is a 7-item instrument that measures the degree to which people perceive they can control factors that influences their lives (i.e., sense of mastery).
Change in sense of societal belonging | Baseline, 9 months (area of Nieuwegein) or 7 months (area of Nijmegen)
  Sense of societal belonging measures how strongly participants feel part of society on an 11-point Likert scale, ranging from 0 to 10. A higher score indicates a stronger sense of societal belonging.
Change in score on Multidimensional Scale of Perceived Social Support (MSPSS) | Baseline, 9 months (area of Nieuwegein) or 7 months (area of Nijmegen)
  The MSPSS is a 12-item instrument that measures social support from (1) family, (2) friends, and (3) a significant other.
Change in social participation | Baseline, 9 months (area of Nieuwegein) or 7 months (area of Nijmegen)
  Social participation measures whether participants engage in daily activities such as paid employment, volunteer work, education and caregiving.
Change in care needs | Baseline, 9 months (area of Nieuwegein) or 7 months (area of Nijmegen)
  Care needs are measured on several domains, including housing & daily life, finances & daily activities, physical & mental health, and social relationships. For each domain, participants were asked to indicate whether they wanted help, whether they received help (and if yes, from whom), and whether this was the right help.

CONTACTS AND LOCATIONS:
Overall Officials: Judith Wolf, PhD, Principal Investigator — Impuls - Netherlands Center for Social Care Research, Radboudumc
Locations (1):
- Radboud university medical center, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No
This study examines vulnerable individuals living in persistent poverty. As the IPD contain sensitive information and publishing these data may deter potential participants, IPD will not be shared with other researchers.